CLINICAL TRIAL: NCT04745364
Title: Mindful Kala: Investigating the Psychosocial Effects of a 4-Week Virtual Bharatanatyam Intervention for Students
Brief Title: Mindful Kala: Virtual Bharatanatyam Wellness Program for Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000029766
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Quality of Life; Cultural Competence; Stress

STUDY DESIGN:
Intervention Model Description: This study uses a waitlist control design. The "call for participants" will be included in the Good Life Center newsletters sent the week of February 8th (if possible) and February 15th. Students will register by 11:59 pm on Friday, February 19th . If they are eligible, within the registration survey, participants will then progress to baseline assessments of stress, well-being, mindful awareness, cultural competence, and feelings of connectedness to the Yale community. Participants will be randomly assigned to either Session One or Session Two.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Session One (Experimental): Session One participants undergo the 4-week course from 2/21/2021 to 3/15/2021
  Interventions: Behavioral: A 4-week Bharatanatyam course from the organization Mindful Kala
- Session Two (Experimental): Session Two participants undergo the 4-week course from 3/22/2021 to 4/12/2021
  Interventions: Behavioral: A 4-week Bharatanatyam course from the organization Mindful Kala

INTERVENTIONS:
Behavioral: A 4-week Bharatanatyam course from the organization Mindful Kala — The 4-week Mindful Kala program focuses on three components of Bharatanatyam: nritta (i.e. technical movements), natya (i.e. storytelling), and nritya (i.e. a combination of movements and narration; nritta + natya).

SUMMARY:
In the current study, the researchers propose to develop and pilot test a Bharatanatyam (i.e. Indian classical dance) program called Mindful Kala with the hopes of decreasing stress and increasing psychosocial well-being, mindfulness, cultural competence, and connectedness amongst a group of college students. The investigators hope that this program can help students cultivate well-being during the challenging and stressful time of COVID-19.

DETAILED DESCRIPTION:
Objectives:

1. Evaluate the effects of the Mindful Kala program on outcomes of health-related measures such as mindfulness, stress, connectedness, and wellbeing amongst students. The investigators hypothesize that participants will experience fewer symptoms of stress, increased mindfulness, increased well-being, and increased connectedness.
2. Evaluate the effects of the Mindful Kala program on changes in measures of cultural competence. The investigators hypothesize that the level of cultural competence will increase among the students.
3. Develop and examine the feasibility and acceptability of a 4-week Mindful Kala program for college students.

ELIGIBILITY:
Inclusion Criteria:

* Yale student
* 18 years of age or older
* Must complete all survey measures
* Is available for all of the designated Session One & Session Two dates and times
* Attends all of the designated Session One & Session Two dates and times

Exclusion Criteria:

* Not a Yale student
* Not 18 years of age or older
* Does not complete all survey measures
* Is not available for all of the designated Session One & Session Two dates and times
* Does not attend all of the designated Session One & Session Two dates and times

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Change in stress from Mindful Kala Intervention | Baseline, 4 weeks
  A primary objective of this study is to determine whether the Mindful Kala program reduces student stress levels. This will be measured by the Perceived Stress Scale (min = 0; max = 4) which consists of 10 scale items. The higher the score, the more likely participants are stressed. Participants who received the intervention in Session One will be compared to the control (Session Two).
Change in subjective well-being from Mindful Kala Intervention | Baseline, 4 weeks
  A primary objective of this study is to determine whether the Mindful Kala program increases subjective well-being. This will be measured by the PERMA Scale (min = 0; max = 10) which consists of 15 scale items. The higher the score, the higher participant well-being. Participants who received the intervention in Session One will be compared to the control (Session Two).
Change in mindful awareness from Mindful Kala Intervention | Baseline, 4 weeks
  A primary objective of this study is to determine whether the Mindful Kala program increases mindful awareness of the present moment. This will be measured by the State Mindfulness Scale for Physical Activity (min = 0; max = 4) which consists of 11 scale items. The higher the score, the more mindful participants are. Participants who received the intervention in Session One will be compared to the control (Session Two).
Change in cultural competence from Mindful Kala Intervention | Baseline, 4 weeks
  A primary objective of this study is to determine whether the Mindful Kala program increases cultural competence. This will be measured by the Cultural Competencies Self-Assessment Survey (min = 0; max = 5) which consists of 26 scale items. The higher the score, the more culturally competent participants are. Participants who received the intervention in Session One will be compared to the control (Session Two).
Change in connectedness from Mindful Kala Intervention | Baseline, 4 weeks
  A primary objective of this study is to determine whether the Mindful Kala program increases connectedness. This will be measured by one question asking questions how connected they feel to the Yale community (min = 1; max = 5). The higher the score, the more connected participants feel. Participants who received the intervention in Session One will be compared to the control (Session Two).

SECONDARY OUTCOMES:
Longitudinal Impact of Mindful Kala on Stress | Baseline, 4 weeks, 8 weeks
  A secondary objective of this study is to determine whether the Mindful Kala intervention resulted in a longitudinal decrease in stress for Session One participants. This outcome is measured by the Perceived Stress Scale (min = 0; max = 4) which consists of 10 scale items. The higher the score, the more stressed participants are.
Longitudinal Impact of Mindful Kala on Well-Being | Baseline, 4 weeks, 8 weeks
  A secondary objective of this study is to determine whether the Mindful Kala intervention resulted in a longitudinal increase in well-being for Session One participants. This outcome is measured by the PERMA Scale (min = 0; max = 10) which consists of 15 scale items. The higher the score, the higher well-being participants have.
Longitudinal Impact of Mindful Kala on Mindfulness | Baseline, 4 weeks, 8 weeks
  A secondary objective of this study is to determine whether the Mindful Kala intervention resulted in a longitudinal increase in mindfulness for Session One participants. This outcome is measured by the Mindfulness Scale for Physical Activity (min = 0; max = 4) which consists of 11 scale items. The higher the score, the more mindful participants are.
Longitudinal Impact of Mindful Kala on Cultural Competence | Baseline, 4 weeks, 8 weeks
  A secondary objective of this study is to determine whether the Mindful Kala intervention resulted in a longitudinal increase in cultural competence for Session One participants. This outcome is measured by the Cultural Competencies Self-Assessment Survey (min = 0; max = 5) which consists of 26 scale items. The higher the score, the more culturally competent participants are.
Longitudinal Impact of Mindful Kala on Connectedness | Baseline, 4 weeks, 8 weeks
  A secondary objective of this study is to determine whether the Mindful Kala intervention resulted in a longitudinal increase in connectedness for Session One participants. This outcome is measured by one question asking questions how connected they feel to the Yale community (min = 1; max = 5). The higher the score, the more connected participants feel.

OTHER OUTCOMES:
Feasibility & Acceptability of Mindful Kala | 8 weeks
  A tertiary objective of this study is to determine the feasibility & acceptability of the Mindful Kala program for college students. This will be measured by asking participants the Feasibility & Acceptability scale (min = 1; max = 5) which consists of 2 scale items, 2 open-ended questions, and 4 multiple choice questions. The higher the score on the scale items, the more participants enjoyed their experience in the Mindful Kala program and the more likely they are to practice Bharatanatyam on their own.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Santos, Doctorate, Principal Investigator — Yale University; Elizabeth Goldfarb, Doctorate, Principal Investigator — Yale University
Locations (1):
- Good Life Center, Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalsa SB, Butzer B. Yoga in school settings: a research review. Ann N Y Acad Sci. 2016 Jun;1373(1):45-55. doi: 10.1111/nyas.13025. Epub 2016 Feb 25. PMID 26919395
- [Background] Koch SC, Riege RFF, Tisborn K, Biondo J, Martin L, Beelmann A. Effects of Dance Movement Therapy and Dance on Health-Related Psychological Outcomes. A Meta-Analysis Update. Front Psychol. 2019 Aug 20;10:1806. doi: 10.3389/fpsyg.2019.01806. eCollection 2019. PMID 31481910
- [Background] Son C, Hegde S, Smith A, Wang X, Sasangohar F. Effects of COVID-19 on College Students' Mental Health in the United States: Interview Survey Study. J Med Internet Res. 2020 Sep 3;22(9):e21279. doi: 10.2196/21279. PMID 32805704
- [Background] Tavormina R, Tavormina MGM. Overcoming Depression with Dance Movement Therapy: A Case Report. Psychiatr Danub. 2018 Nov;30(Suppl 7):515-520. PMID 30439838
- [Background] Misra S, Le PD, Goldmann E, Yang LH. Psychological impact of anti-Asian stigma due to the COVID-19 pandemic: A call for research, practice, and policy responses. Psychol Trauma. 2020 Jul;12(5):461-464. doi: 10.1037/tra0000821. Epub 2020 Jun 11. PMID 32525390
- See also: Related Info — http://www.apa.org/news/press/releases/2014/02/teen-stress
- See also: Related Info — http://dancesinthefarsouth.weebly.com/information/3-components-of-bharatnatyam
- See also: Related Info — http://www.apa.org/helpcenter/stress-body